CLINICAL TRIAL: NCT04810780
Title: Safety and Efficacy of DUO Extended Set: Combined Glucose Sensor and Infusion Set.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Prof. Amir Tirosh, Director, Division of Endocrinology, Sheba Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Sheba-20-7386-at-ctil
Record Dates: First submitted 2021-03-21; First posted 2021-03-23 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 1st arm (Experimental): Wearing the Duo infusion set for up to 1 month or up to 4 infusion set failures.
  Interventions: Device: DUO Extended Set

INTERVENTIONS:
Device: DUO Extended Set — to evaluate saftey and efficacy of DUO extended set combined with glucose sensor

SUMMARY:
The study will follow subjects for 28 days while using an DUO extended infusion set combined with glucose sensor. the objective is to evaluate saftey and efficacy of the set in adult patient with type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of type 1 diabetes for at least one year
2. Using a MiniMed™ 670G or 640G Insulin pump with Guardian sensor
3. Age 18 to 80 years
4. Hemoglobin A1c level less than or equal to 10%
5. Not currently known to be pregnant, nor planning pregnancy during the study.
6. Willingness to follow the protocol and sign the informed consent

Exclusion Criteria:

1. A known medical condition that in the judgment of the investigator might interfere with the completion of the protocol.
2. Pregnant or lactating females
3. Subject has Glycosylated hemoglobin (HbA1c) > 10 % at time of screening.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Primery Effectivness Endpoint | 28 days
  Precent of catheters reaching 7- day without set failure.

CONTACTS AND LOCATIONS:
Overall Officials: amir Tirosh, MD PhD, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Tel Litwinsky, Israel

IPD SHARING:
Plan to Share IPD: No